CLINICAL TRIAL: NCT00840723
Title: Bronchoscopy-Assisted Sampling of Cells and Fluid From the Lower Respiratory Tract of Human Subjects
Brief Title: Bronchoscopy Assisted Sampling of Cells and Fluid From the Lower Respiratory Tract of Human Subjects
Acronym: SCCOR Bronch
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Raymond Coakley, MD, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Other Study IDs: CTRC 2799; NHLBI P50-HL084934
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Respiratory Diseases
Keywords: Healthy smokers; Current cigarette smokers; No lung disease
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, Bronchial Lavage Fluid (BALF), cytology brushings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Current smokers: Current cigarette smokers with no other illness
- Healthy controls: Healthy non smokers

SUMMARY:
The purpose of this research study is to collect cells and liquid from the air passages of healthy adults, both smokers and non-smokers. These samples will be used for test-tube studies to explore mechanisms of diseases of the respiratory tract, and to compare the samples between people who smoke cigarettes and people who don't. Obtaining these samples requires an invasive procedure called "bronchoscopy".

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers
* Must be otherwise healthy with no chronic illness

Exclusion Criteria:

* Asthma
* Smoking related lung disease (including bronchitis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current cigarette smokers who are otherwise healthy (no lung disease or other chronic illness and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The goal of this project is to define the effect of smoking on key aspects of airway biology. These studies will also provide crucial & novel definition of airway biology in smokers against which COPD & CF patients will be compared. | At the time of bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Coakley, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States